CLINICAL TRIAL: NCT04634175
Title: Yoga Intervention Practice as a Complementary and Integrative Treatment for Compulsive Sexual Behavior Disorder: Randomized Controlled Trial
Brief Title: Yoga Intervention for Compulsive Sexual Behavior Disorder
Acronym: CSBD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30117919.5.0000.0068
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Compulsive Sexual Behavior
Keywords: Sexual Compulsion; Hypersexuality; Sex addiction; Disorder
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder; Disease

STUDY DESIGN:
Intervention Model Description: Pre-test-post-test.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Volunteers, health care professionals and researchers will not have access to randomization and will also not know which intervention group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga group (Experimental): The yoga group will practice yoga intervention.
  Interventions: Behavioral: Yoga intervention
- Sham group (Active Comparator): The sham group will practice muscle stretching intervention.
  Interventions: Behavioral: Sham intervention

INTERVENTIONS:
Behavioral: Yoga intervention — The yoga intervention is composed of kundalini yoga techniques.
  Arms: Yoga group
Behavioral: Sham intervention — The sham intervention is composed of stretching and muscle flexion techniques.
  Arms: Sham group

SUMMARY:
Yoga intervention as a complementary and integrative treatment for compulsive sexual behavior disorder (CSBD).

The hypothesis is that participants with CSBD, after being submitted to the protocol of the yoga intervention group in relation to those submitted to the intervention protocol Shan of the control group, present less severe sexual compulsiveness.

DETAILED DESCRIPTION:
Yoga intervention practice as a complementary and integrative treatment for compulsive sexual behavior disorder (CSBD), a randomized clinical trial, in a sample of male individuals who spontaneously seek treatment at the Psychiatry Institute of Hospital das Clínicas, University of São Paulo.

The volunteers with CSBD will be randomized by statistical software in two groups, yoga intervention practice and Shan intervention practice, to participate in a twelve-week program of daily practices of the mind-body practices protocol.

The participants will be evaluated by measuring instruments at time 1 (4th week), time 2 (8th week) and time 3 (12th week).

The primary objective of the study is to investigate the effectiveness of yoga intervention practice in decreasing the symptoms (sexual compulsiveness) of the CSBD.

The secondary objectives of the study are to investigate the effectiveness of the yoga intervention practice in reducing the severity of impulsivity, hypersexuality, anxiety, depression, improving the level of quality of life, and increasing adherence to total treatment.

ELIGIBILITY:
Inclusion Criteria:

1. They must have a minimum score of 28 on the Sexual Compulsiveness Scale (range 10 - 40) or a minimum score of 20 on the Screening Inventory of Hypersexual Disorder (range 0 - 28) and a minimum score of 14 on the Beck Anxiety Inventory (range of 0 - 63);
2. Male;
3. Being Brazilian;
4. Literate in Brazilian Portuguese;
5. Have a satisfactory cognitive level to understand and respond to self-responsive inventories;
6. Have availability to participate in a daily mind-body Intervention program for 12 weeks.

Exclusion Criteria:

1. Individuals who meeting the criteria for Substance-Related Disorder and Addictive Disorders (DSM-5, 483);
2. Individuals who meeting the criteria for Paraphilic Disorders (DSM-5, 685);
3. Individuals who meeting the criteria for Gender Dysphoria (DSM-5, 451);
4. Individuals who meeting the criteria for Spectrum of Schizophrenia and other Psychotic Disorders (DSM-5, 87);
5. Individuals who meeting the criteria for Hypomanic or Manic Episode of Mood Disorder (DSM-5, 123);
6. Individuals who meeting the criteria for Neurocognitive Disorders (DSM-5, 591);
7. Individuals who meeting the criteria for Other Mental Disorders (DSM-5, 707);
8. Individuals who have already have practiced kundalini yoga;
9. Individuals who use psychiatric medication and cannot maintain the stability and regularity of the dosage three months before and during the intervention program;
10. Individuals who have attended psychotherapy in the last six months in weekly sessions and with at least 75% attendance;
11. Individuals who have significant spinal problems and / or physical limitations that may interfere with yoga practice, for example, overweight, severe lung and / or cardiovascular disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Sexual Compulsivity Scale (SCS) | Baseline, 4th week, 8th week and 12th week
  Changes in the total score of Sexual Compulsivity Scale, the scores vary between 10 and 40, with the highest ones indicating greater sexual compulsiveness.

SECONDARY OUTCOMES:
Barrat Impulsivity Scale (BIS 11) | Baseline, 4th week, 8th week and 12th week
  Changes in the total score of Barrat Impulsivity Scale, the scores vary between 1 and 30, with the highest ones indicating greater impulsivity.
Hypersexual Disorder Screening Inventory (HDSI) | Baseline, 4th week, 8th week and 12th week
  Changes in the total score of Hypersexual Disorder Screening Inventory score, the scores vary between 0 and 28, with the highest ones indicating greater hypersexuality.
Beck Anxiety Inventory (BAI) | Baseline, 4th week, 8th week and 12th week
  Changes in the total score of Beck Anxiety Inventory, the scores vary between 0 and 63, with the highest ones indicating greater anxiety.
Beck Depression Inventory (BDI) | Baseline, 4th week, 8th week and 12th week
  Changes in the total score of Beck Depression Inventory, the scores vary between 0 and 63, with the highest ones meaning greater depression.
World Health Organization Quality of Life (WHOQOL-bref) | Baseline and 12th week
  Changes in the total score of World Health Organization Quality of Life-bref, the scores vary from 26 to 130, with the highest ones meaning greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Scanavino, PHD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Instituto de Psiquiatria do Hospital das Clínicas da Universidade de São Paulo[University of Sao Paulo General Hospital], São Paulo, São Paulo, Brazil